CLINICAL TRIAL: NCT03739476
Title: Controlled, Double-blind, Randomized Clinical Trial for Prophylaxis of Postoperative Delirium in High Risk Surgical Patients With Quetiapine
Brief Title: Clinical Trial With Quetiapine Prophylaxis Postoperative Delirium in High Risk Surgical Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the crisis SARS-COV-2 pandemic: recruitment of patients for the trial is stopped, healthcare pressure generated, suspend the non-essential scheduled surgical activity and on June 30, 2020 medication expired, funding has been exhausted.
Sponsor: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other); Grupo Español de Rehabilitación Multimodal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QUEPRO; GRS1855/A/18 (Other Grant/Funding Number: Gerencia Regional de Salud de Castilla y León-JCYL); 17/1358 (Other: IBSAL (INSTITUTO DE INVESTIGACION BIOMEDICA DE SALAMANCA); 2016-004117-27 (EudraCT Number)
Record Dates: First submitted 2018-10-18; First posted 2018-11-13 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Delirium
Keywords: Postoperative; Delirium; Quetiapine; Prophylaxis
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Intervention Model Description: one arm treatment. one arm placebo.
Who Masked: Participant, Investigator
Masking Description: double blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Quetiapine 25 milligrams 1 hour after surgery and each 12 hours for 3 days
  Interventions: Drug: Quetiapine 25 milligrams capsule
- control (Placebo Comparator): Placebo 1 hour after surgery and each 12 hours for 3 days
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Quetiapine 25 milligrams capsule — Compare the incidence of postoperative delirium.
  Other Names: Experimental arm
  Arms: Interventional
Drug: Placebo oral capsule — Compare the incidence of postoperative delirium.
  Other Names: Control arm
  Arms: control

SUMMARY:
Double blinded Clinical trial to test efficacy of Quetiapine versus placebo in reducing postoperative delirium in high risk surgical patients after three days of treatment.

DETAILED DESCRIPTION:
This study evaluates postoperative delirium in high risk surgical patients to know the incidence of postoperative delirium in patients at risk, over 65 years, treated early with prophylactic quetiapine versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 65 years-old patients who will be undergoing major surgery (noncardiac) and having an equal or greater score of 5 on the scale Delphi.
* Age: 70-79 years: 1 point; ≥80 years: 2 points.
* Physical activity: need for assistance, not self-sufficient: 2 point.
* Alcoholism: 1 point.
* Hearing Impaired: 1 point.
* History of delirium: 2 points.
* Emergency surgery: 1 point.
* No laparoscopic surgery: 2 points.
* Admission critical Units: 3 points.
* Value of C-reactive protein (CRP) ≥ 10 milligrams (mg) / decilitre (dL): 1 point

Exclusion Criteria:

* Allergy to quetiapine.
* Patients with a score less than 5 on the Delphi scale.
* Diagnosis of delirium at admission.
* Cardiological diseases: corrected QT interval (QTc) ≥ 460 millisecond (msec) in men, ≥ 470 msec in women, recent myocardial infarction or cardiac decompensation, 2-3° degree atrioventricular block or history of torsades de pointes arrhythmias or ventricular arrhythmias, bradycardia...
* Hypokalemia ≤ 3 milliequivalent (mEq) / Potassium chloride (KCl).
* History of drug use.
* Patients on Antipsychotic or antidopaminergic treatment (chlorpromazine, clozapine, olanzapine, risperidone, haloperidol, quetiapine, paliperidone, amisulpride).
* Parkinson's disease.
* Test MINIMENTAL ≤ 24.
* Corps or vascular dementia Levi.
* Hypokinetic movement disorder.
* History of neuroleptic malignant syndrome.
* Central Anticholinergic Syndrome.
* Epilepsy.
* Patients with a wight less than 50 or greater than 200 kg (kilograms).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
To Know the incidence of postoperative delirium in patients at risk, over 65 years, treated early with prophylactic quetiapine versus placebo. | 28 (± 2) days from the start of treatment in each patient.
  Proportion of patients diagnosed with delirium (number of cases of delirium / total number of patients) within the first four days in both arms.
  65 years, treated early with prophylactic quetiapine versus placebo.

SECONDARY OUTCOMES:
Days without delirium, if it appears. | 28 ± 2 days from the start (first dose) of treatment with quetiapine.
  Number of days from the start of treatment until delirium.
Duration of delirium, if it appears. | 28 ± 2 days from the start (first dose) of treatment with quetiapine.
  Number of days with delirium, if it appears. Perceived quality of life.
  Mortality (all causes).
Severity of delirium measured with a validated scale. time of appearance the duration and severity. use of another antipsychotics. | 28 ± 2 days from the start (first dose) of treatment with quetiapine.
  Severity of delirium measured with a the Delirium Rating Scale-Revised-98 (DRS-R-98).
Dose of other antipsychotic (haloperidol). | 28 ± 2 days from the start (first dose) of treatment with quetiapine.
  Total dose (mg) of other antipsychotic to control symptoms of delirium.
Degree of sedation. | 28 ± 2 days from the start (first dose) of treatment with quetiapine.
  Degree of sedation measured with a validated scale Richmond Agitation-Sedation Scale (RASS).
Measurement of corrected QT interval (QTc) prolongation. | 28 ± 2 days from the start (first dose) of treatment with quetiapine.
  Increased (msec) ECG control.
Evaluation of extrapyramidal symptoms. | 28 ± 2 days from the start (first dose) of treatment with quetiapine.
  Presence o absence of extrapyramidal symptoms (tremor, involuntary movements, rigidity).
Days in hospital from surgery. | 28 ± 2 days from the start (first dose) of treatment with quetiapine.
  Number of days from surgery until discharge.
Perceived general well-being. | 28 ± 2 days from the start (first dose) of treatment with quetiapine.
  Evaluation of quality of life using Short Form-36 Health Survey questionnaire (SF36).
Mortality (all causes) | 28 ± 2 days from the start (first dose) of treatment with quetiapine.
  Mortality at discharge and at 28 (± 2) days before the start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Sanchez-Barrado, MD, Principal Investigator — Investigator
Locations (1):
- Complejo Asistencial Universitario de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT03739476/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT03739476/ICF_001.pdf